CLINICAL TRIAL: NCT00481273
Title: AVIDA The Vidaza® (Azacitidine) Patient Registry
Acronym: AVIDA
Status: Completed | Type: Observational
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: AVIDA
Record Dates: First submitted 2007-05-30; First posted 2007-06-01 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Myelodysplastic Syndromes
Keywords: MDS
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Azacitidine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Azacitidine — Physician's discretion
  Other Names: Vidaza(R)

SUMMARY:
This registry is a prospective, multi-center, observational study compiling data on the natural history and management of patients receiving Vidaza, and will provide unique insights into the management of myelodysplastic syndromes (MDS) and other hematological disorders and the impact of these disorders on patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient who is deemed appropriate for treatment with Vidaza® by his or her clinician, but who has not already started receiving Vidaza® treatment.
* Patient who is able to read and speak English.
* Patient who is willing and able to provide informed consent.
* Patient who agrees to complete patient assessment questionnaires.

Exclusion Criteria:

* Patients who are currently being treated with Vidaza®.
* Patients who are concurrently participating in a clinical trial.
* Patients unwilling or unable to complete the baseline and follow-up questionnaires.
* Patients who are deemed inappropriate for treatment with Vidaza®.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Community-based hematology/oncology centers
Sampling Method: Probability Sample
Enrollment: 479 (Actual)
Dates: Start 2006-10-31 (Actual); Primary Completion 2010-08-31 (Actual); Study Completion 2010-08-31 (Actual)

PRIMARY OUTCOMES:
Vidaza usage | Approximately 4 years
  Describe current usage patterns for Vidaza in the community
Concomitant care and treatment | Approximately 4 years
  Document common concomitant care procedures and treatments used in conjnction wtih Vidaza
Duration and number of cycles | Approximately 4 years
  Correlate duration and number of Vidaza treatment cycles with clinical response as defined by 2006 International Working Group for Myeleodysplastic Syndrome
Publication | Approximately 4 years
  Produce publications to support further clinical development and disseminate information on treatment best practices

CONTACTS AND LOCATIONS:
Overall Officials: David L. Grinblatt, MD, Principal Investigator — Endeavor Health
Locations (1):
- AVIDA Registry Help, Kansas City, Missouri, United States

REFERENCES:
- [Background] Grinblatt DL, Sekeres MA, Komrokji RS, Swern AS, Sullivan KA, Narang M. Patients with myelodysplastic syndromes treated with azacitidine in clinical practice: the AVIDA registry. Leuk Lymphoma. 2015 Apr;56(4):887-95. doi: 10.3109/10428194.2014.935366. Epub 2014 Aug 20. PMID 24956145